CLINICAL TRIAL: NCT04617301
Title: Three-dimensional Volumetric/ Linear Analysis and Axial Classification of Root Resorptions Using Cone Beam Computed Tomography: A Retrospective Study
Brief Title: Volumetric Analysis of Resorption Types on CBCT
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2020/98
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Endodontic Disease; Tooth Resorption
Keywords: cone beam computed tomography; endodontics; tooth Resorption
MeSH Terms: conditions — Dental Pulp Diseases; Tooth Resorption

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1. Internal root resorption (IRR): Internal root resorption is the progressive destruction of intraradicular dentin and dentinal tubules along the middle and apical thirds of the canal walls as a result of clastic activities. It is seen as a radiolucent area around the pulpal cavity, usually of incisors and mandibular molars. The various etiological factors suggested for internal root resorption include traumatic injury; infection and orthodontic treatment.
- Group 2. external cervical resorption (ECR): Cementum is considered to protect the underlying root dentin from being resorbed. It is broadly accepted that damage to or deficiency of this protective cementum layer below the epithelial attachment exposes the root surface to osteoclasts, which then resorb the dentin.
  Clinical sign; Located in cervical region of tooth Pink spot might be noted by patient/dentist Tooth usually responds positively to vitality tests unless there is pulpal involvement (in very advanced cases) Spontaneous and profuse bleeding on probing Sharp, thinned out edges around the resorptive cavity
- Grup 3. external replacement resorption (ERR): external replacement resorption also known as trauma-induced resorption - and this resorption may occur in teeth that also have external inflammatory resorption. This review will not discuss external replacement resorption in detail but it will be mentioned where relevant as both types of resorption may occur in some cases. This is because replacement resorption is a consequence of the same injuries that typically cause external inflammatory resorption - such as intrusion and avulsion where there is significant damage to the external root surface during the injury, as well as sometimes during the repositioning/ replantation of the tooth.

SUMMARY:
More accurate management of resorption can be achieved thanks to the three-dimensions volumetric and linear analysis, and the axial classification presented in this study.

DETAILED DESCRIPTION:
The aim of this study was to investigate the volumetric and linear analysis, and to present the axial classification of root resorptions using cone beam computed tomography (CBCT).

A total of 43 teeth of external cervical resorption (ECR) (n=27), external replacement resorption (ERR) (n=4) and internal root resorption (IRR) (n=12) were identified from 34 patients. The volume of resorption and total tooth, the widest lengths of these resorptions, and the amount of thinnest dentin thickness around them were measured and compared according to age and sex. Additionally, the eight regional axial classification was performed and the percentages in these regions were evaluated. Significance was set at p=0.05 for statistical analysis.

More accurate management of resorption can be achieved thanks to the three-dimensions volumetric and linear analysis, and the axial classification presented in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cases of resorption that had CBCT images

Exclusion Criteria:

* those presenting pathologic lesions, congenital/developmental anomalies or teeth with root canal filling
* those whose CBCT scans failed to present satisfactory quality.
* Additionally, SR, TAP, and EIR cases were excluded because their true dimensions could not be completely determined before resorption.

Ages: 12 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases of resorption that had CBCT images were included in the study. Radiographic features of resorption were defined in the images of 34 patients in accordance with these criteria. A total of 43 teeth with ECR (n=27), ERR (n=4), and IRR (n=12) were identified from 34 patients.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Volume of total tooth and resorbed area | for three months from the beginning of the study
  The total volume and the resorption volume were measured with used 3D semi-automatic segmentation program (ITK-SNAP 2.4)
Measurement widest mesio-distal length, bucco-lingual length and corono-apical length of the resorbed lesion | for three months from the beginning of the study
  Linear measurement were measured with used Planmeca ProMax 3D Classic (Planmeca Promax 3D; Planmeca Oy; Helsinki, Finland)
Linear measurements for thinnest dentin (buccal, distal, mesial and lingual/ palatinal) and resorbed area (mesio-distal length and bucco-lingual length) were made on axial sections | for three months from the beginning of the study
  Linear measurement were measured with used Planmeca ProMax 3D Classic (Planmeca Promax 3D; Planmeca Oy; Helsinki, Finland)
The corono-apical length was measured on sagittal sections where the tooth axis was perpendicular to the ground plane. | for three months from the beginning of the study
  Linear measurement were measured with used Planmeca ProMax 3D Classic (Planmeca Promax 3D; Planmeca Oy; Helsinki, Finland)
the axial section of the tooth was divided into eight parts and regional settlement classification was performed | for three months from the beginning of the study
  Segmentation were made with used Planmeca ProMax 3D Classic (Planmeca Promax 3D; Planmeca Oy; Helsinki, Finland)

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Nil Günaçar, Study Chair — Recep Tayyip Erdogan University Training and Research Hospital
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

REFERENCES:
- [Background] Heithersay GS. Clinical, radiologic, and histopathologic features of invasive cervical resorption. Quintessence Int. 1999 Jan;30(1):27-37. PMID 10323156
- [Background] Patel S, Dawood A, Wilson R, Horner K, Mannocci F. The detection and management of root resorption lesions using intraoral radiography and cone beam computed tomography - an in vivo investigation. Int Endod J. 2009 Sep;42(9):831-8. doi: 10.1111/j.1365-2591.2009.01592.x. Epub 2009 Jul 14. PMID 19627378